CLINICAL TRIAL: NCT06677450
Title: Effectiveness of Pain Neuroscience Education in Rotator Cuff Related Shoulder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Büşra Aksan Sadıkoğlu, MSc, PT, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IUC2025
Record Dates: First submitted 2024-10-31; First posted 2024-11-06 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Rotator Cuff Related Shoulder Pain; Impingement Syndrome; Shoulder Tendinopathy
Keywords: shoulder; pain; rotator cuff tear; pain neuroscience
MeSH Terms: conditions — Pain; Rotator Cuff Injuries | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Active Comparator): Exercise program
  Interventions: Other: Exercise
- Pain Neuroscience Education Group (Experimental): Pain neurosicence education with exercise program
  Interventions: Other: Pain neuoroscience education; Other: Exercise

INTERVENTIONS:
Other: Pain neuoroscience education — Pain neurosicence education will be applied 1 day / 6 weeks at the beginning of one of the weekly exercise sessions in addition to the exercise program. The educations will include the definition and general characteristics of pain, pain physiology, peripheral neuropathic pain, the role of the brain in pain perception, tissue healing, peripheral and central sensitization, the effects of emotional, psychological and social factors on the pain process and pain coping strategies.
  Arms: Pain Neuroscience Education Group
Other: Exercise — Exercise program will be applied 2 days/week for 6 weeks and will consist of 3-phase stretching and motor control/progressive resistance exercises.
  Arms: Exercise Group
Other: Exercise — Exercise program will be applied 2 days/week for 6 weeks and will consist of 3-phase stretching and motor control/progressive resistance exercises.
  Arms: Pain Neuroscience Education Group

SUMMARY:
The aim of this randomized controlled trial was to investigate the effects of pain neuroscience education added to exercise on pain intensity, disability, pain threshold, pain catastrophizing, pain beliefs, pain knowledge, and quality of life in rotator cuff related shoulder pain.

DETAILED DESCRIPTION:
Shoulder pain associated with rotator cuff injuries is a common clinical condition, with a global prevalence of 20.7%. Its etiology is multifaceted, and it is often reported that pain does not align with findings from diagnostic imaging. Recent studies have indicated that psychological factors, such as central sensitization and pain beliefs, play a significant role in patients with shoulder pain. Although exercise is recommended as the first-line treatment, approximately 50% of patients return with persistent pain complaints 6 to 12 months later. Treatments focused on the local tissue pathology-pain model are inadequate in addressing more complex and chronic pain issues related to central sensitization and neuroplasticity. There is a need for an approach that aims to desensitize the nervous system by focusing on neurophysiology and the representation and meaning of pain, rather than a traditional biomedical model.

Pain neuroscience education is a treatment strategy that offers patients the opportunity to reconceptualize their ideas about pain, thereby changing negative beliefs and misconceptions regarding it. Recent literature has provided strong evidence that pain neuroscience education can alter pain intensity, pain knowledge, disability, and pain behaviors in patients with musculoskeletal pain. However, studies investigating patients' perceptions of pain neuroscience education in relation to rotator cuff related shoulder pain and the feasibility of implementing such education have emerged. Despite the limited existing evidence, the efficacy of pain neuroscience education combined with exercise for individuals with rotator cuff related shoulder pain has not been supported by a randomized controlled trial, indicating a need for further research in this area.

Therefore, the aim of this study is to investigate the effects of pain neuroscience education, applied in addition to exercise, on pain intensity, disability, pain threshold, pain catastrophizing, pain beliefs, pain knowledge, and quality of life in individuals with rotator cuff related shoulder pain.

Patients with rotator cuff related shoulder pain the ages of 40 and 65 will be randomly divided into two groups: Group 1 (pain neuroscience education + exercise) and Group 2 (exercise). Interventions will be applied for 12 sessions (twice a week for 6 weeks). The patients will be assessed at baseline and at the end of the 6-week intervention.

After the demographic and clinical characteristics of the patients were evaluated with the demographic information form, pain intensity will be evaluated with the Numerical Pain Rating Scale (NPRS), disability with the Shoulder Pain and Disability Index (SPADI), pressure pain threshold with the Algometer, pain catastrophizing with the Pain Catastrophizing Scale, pain beliefs with the Pain Beliefs Scale, change in pain knowledge with the Revised Pain Neurophysiology Scale, quality of life with the Short Form-12 (SF-12), and patient satisfaction with the Global Change Rating Scale.

ELIGIBILITY:
Inclusion Criteria:

* Being aged between 40 and 65 years
* Presence of shoulder pain for at least 3 months
* At least one positive finding in each of the following categories; 1) Painful arc finding during flexion or abduction, 2) Positive Neer's or Kennedy-Hawkins Tests, 3) Pain with resisted external rotation, abduction or empty can test
* Pain level of at least 3 and at most 7 according to Visual Analogue Scale (VAS) at rest
* Being literate

Exclusion Criteria:

* Systemic inflammatory shoulder pain
* Having had a shoulder dislocation or fracture in the last 12 months
* Having had a shoulder surgery
* Having received physiotherapy or corticosteroid injection treatment for the shoulder in the last 3 months
* Presence of adhesive capsulitis (passive shoulder ROM <50%)
* Presence of vision and hearing problems
* Having been diagnosed a disease that may cause neurological-cognitive changes and prevents understanding the content of the ANE program

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | At the baseline and end of 6-week intervention
  The Numeric Pain Rating Scale (NPRS) will be used to evaluates pain levels. In the NPRS, participants are asked to verbally rate the intensity of their pain on a scale from 0 to 10.
Disability | At the baseline and end of 6-week intervention
  The disability level of individuals will be measured with the Shoulder Pain and Disability Index (SPADI). SPADI is a 13-item scale, with 5 items measuring pain and 8 items measuring disability, for a total of 2 subscales to assess the level of perceived disability. The average of the 2 subscales out of 100 is taken for the total score; a higher score indicates greater disability.

SECONDARY OUTCOMES:
Pressure Pain Threshold | At the baseline and end of 6-week intervention
  A mechanical pressure algometer will be used to measure the pressure pain threshold of the muscles around the shoulder. The device consists of a 1 cm2 rubber disc connected to a manometer that displays the values in kg/cm2 (0 to 10 kg). The average of three trials will be calculated, allowing a 30-second rest period between each trial.
Pain Catastrophizing | At the baseline and end of 6-week intervention
  The level of catastrophizing of individuals will be measured with the Pain Catastrophizing Scale. The 5-point scale, consisting of 13 items, assesses destructive thoughts and feelings related to pain. A score of 0 means "never" and a score of 4 means "always". A high score indicates the severity of pain.
Pain Beliefs | At the baseline and end of 6-week intervention
  Individuals' pain beliefs will be measured with the Pain Beliefs Scale. It is a 12-question scale that evaluates organic and psychological belief status regarding the source and outcome of pain. There is an organic beliefs subtest consisting of eight items and a psychological beliefs subtest consisting of four items. Scoring for each item varies between 1-6.
Pain Knowledge | At the baseline and end of 6-week intervention
  Pain knowledge will be measured with the Pain Neurophysiology Questionnaire (Revised-NPQ-TR) scale. It is a 12-item scale that patients can apply themselves and evaluates the level of knowledge about pain neurophysiology. Each item has the answer options "true-false-undecided". The scale is scored out of 12, with 1 point given for each correct answer. 0 points are given for wrong answers and undecided answers.
Health-Related Quality of Life | At the baseline and end of 6-week intervention
  Health-related quality of life will be measured using the SF-12 (Short Form-12). The SF-12 provides two sub-scores: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). The PCS is derived from the sub-dimensions of general health, physical functioning, physical role, and bodily pain, while the MCS is derived from the sub-dimensions of social functioning, emotional role, mental health, and energy.
Patient Satisfaction | End of the 6-week intervention
  Patient Satisfaction will be measured with the Global Rating Scale. It is a commonly used self-reported scale to measure a person's perceived change in health status and consists of a single question, 'How would you describe yourself compared to before treatment?', asking the patient to rate their change with respect to a specific condition over a specified period of time.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No